CLINICAL TRIAL: NCT06348186
Title: Fascial Tissue Response to Manual Therapy: Implications in Long COVID-19
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of the State of Santa Catarina (Other)
Collaborators: Fundação de Amparo à Pesquisa e Inovação do Estado de Santa Catarina (Unknown)
Responsible Party: Principal Investigator, Gilmar Moraes Santos, PT, Associate Professor, University of the State of Santa Catarina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Fascial Tissue Response
Record Dates: First submitted 2024-04-03; First posted 2024-04-04 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-05

CONDITIONS: COVID-19
Keywords: Long COVID; Manual Therapy; Fascia; Rehabilitation
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two or groups, typically an intervention group (fascia-focused manual therapy) and a control group. Participants are randomly allocated. Participants and outcomes assessor are blinded.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Guidebook (Other)
  Interventions: Other: Guidebook
- Guidebook and Myofascial Reorganization® (RMF). (Experimental)
  Interventions: Other: Guidebook and Myofascial Reorganization® (RMF).

INTERVENTIONS:
Other: Guidebook — Folder that will be given to the participant to carry out 5 minutes of intervention daily
  Arms: Guidebook
Other: Guidebook and Myofascial Reorganization® (RMF). — The intervention will be carried out once a week for 30 minutes for 6 weeks. It will include passive, active-assisted moments (with and without load). In addition to a folder that will be given to the participant to carry out 5 minutes of intervention daily.
  Arms: Guidebook and Myofascial Reorganization® (RMF).

SUMMARY:
According to the World Health Organization (WHO), as of mid-September 2022, more than 21 million Brazilians have recovered from COVID-19. However, post-infection symptoms continue to appear months after the end of the acute infection, a syndrome called long COVID. Therefore, the aim of this study is to investigate the responses of fascia-focused manual therapy in participants with long COVID.

DETAILED DESCRIPTION:
Participants reported to have long COVID, of both sexes, aged between 20 and 80 years, from the community, outpatient clinics and hospitals will be evaluated. The treatment of participants will be carried out at the CEFID-UDESC Physiotherapy School Clinic, where they will undergo assessment of the biomechanical and viscoelastic properties of tissues, postural control, pain and quality of life. For normality analysis, the Shapiro-Wilk test will be applied, and according to the distribution of the data, parametric or non-parametric tests will be used. Pre- and post-assessment and treatment data will be compared using descriptive statistics and Student's t-test with a significance level of p=0.05 for parametric data or Wilcoxon for non-parametric data.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with long COVID, of both sexes, aged between 20 and 80 years, from the community, outpatient clinics and hospitals.

Exclusion Criteria:

* Participants with suspected deep vein thrombosis; Participants with neurological disorders.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Functioning and disability | 6 weeks
  Will be assessed using the "World Health Organization Disability Assessment" questionnaire (WHO-DAS 2.0), translated and validated for the Brazilian population by Silveira et al. (2013).
Biomechanical and tissue viscoelastic properties | 6 weeks
  Will be evaluated by MyotonPro (MytonPro, Myoton Ltd.s., Tartu, Estonia)

SECONDARY OUTCOMES:
Work capacity | 6 weeks
  Will be assessed by the "Work Limitations Questionnaire, WLQ-25" translated and validated for the Brazilian population by Soárez et al (2007).
Level of Quality of life | 6 weeks
  Will be assessed by the "World Health Organization Questionnaire" in its short version, validated in the Brazilian population and by the "Medical Outcomes Study 36-Item Short Form Health" questionnaire Survey" validated for Brazilian-Portuguese.
Upper limb dysfunctions | 6 weeks
  Will be assessed using the Arm, Shoulder and Hand Dysfunctions questionnaire (DASH), translated and validated for the Brazilian population by Orfale et al (2005).
Balance | 6 weeks
  Will be assessed using the Neurocom Balance Platform (VRS Sport) and its NeuroCom®Balance Manager program (Neurocom International, Inc, Clackamas, OR).

CONTACTS AND LOCATIONS:
Locations (1):
- Santa Catarina State University, Florianópolis, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: No